CLINICAL TRIAL: NCT02679170
Title: Observational Study to IDEntify Patients With Advanced/Metastatic NSCLC and ALK and ROS1 Translocation and to Establish Their Therapeutic Management (IDEALK&ROS)
Brief Title: Study to IDEntify Patients With Advanced/Metastatic Non Small Cell Lung Cancer (NSCLC) and ALK and ROS1 Translocation and to Establish Their Therapeutic Management (IDEALK&ROS)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8081057; IDEALKROS (Other: Alias Study Number); IDEALK (Other: Alias Study Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-10 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: ALK+, ROS1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Routine clinical practice group (NSCLC ALK+, ROS1): Patients diagnosed and treated following routine clinical practice, for their NSCLC ALK+ or ROS1
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Treatment with crizotinib following routine clinical practice

SUMMARY:
Prospective observational study to IDEntify patients with advanced/metastatic NSCLC and ALK and ROS1 translocation and to establish their therapeutic management (IDEALK&ROS)

ELIGIBILITY:
Inclusion Criteria:

For ALK Incidence substudy

* Patients with Advanced or metastatic non-small cell lung cancer
* Patients who will be screened for anaplastic lymphoma kinase (ALK) rearrangement
* Age > 18 years For ALK treatment substudy (retrospective and prospective)
* Age > 18 years
* Confirmed anaplastic lymphoma kinase (ALK)-positive tumour
* Patients treated with crizotinib under routine clinical practice
* Patients with a minimum data registered at the medical history
* For the patients that will be recruited prospectively: Patients must have a signed informed consent document.

For the ROS1 treatment sub-study (retrospective only):

* Age > 18 years
* Confirmation of NSCLC with ROS1-positive translocation
* Have been eligible to receive treatment with crizotinib according to routine clinical practice since the market launch of the ROS1 indication in Spain on 8 February 2017 until the opening of the site.
* Patients should have a predetermined minimum amount of data recorded in their medical records.

Exclusion Criteria:

* Any patient who does not meet any of the inclusion criteria defined in the previous section, depending on the sub-study for which they are included.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC Patients, ALK +translocation confirmed, ROS1+translocation confirmed
Sampling Method: Non-Probability Sample
Enrollment: 692 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- Spain (32):
  - Hospital Clínico Univ. de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Complejo Hospitalario de Jerez, Jerez de la Frontera, Cadiz
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital General Mancha Centro, Alcázar de San Juan, Ciudad REAL
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Cruces, Barakaldo, Vizcaia
  - Hospital Universitario de Albacete, Albacete
  - Hospital Universitario Clinic i Provincial, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Puerta del Mar, Cádiz, Cadiz
  - Complejo Hospitalario de Jaen, Jaén
  - Complejo Hospitalario Universitario Insular Materno-Infantil, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital Universitario San Pedro, Logroño, Logroño
  - Hospital Universitario Lucus Augusti (HULA_ Lugo), Lugo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jimenez Diaz, Madrid
  - H.U. La Paz, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Ourense (CHUOU), Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - HU Son Llatzer, Palma de Mallorca / Servicio de Oncología Médica, Palma de Mallorca
  - Hospital Universitario de la Candelaria, Tenerife, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen de La Salud, Toledo
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Universitario de Vigo- Hospital Álvaro Cunqueiro / Servicio de Oncología Médica, Vigo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Aguado de la Rosa C, Cruz Castellanos P, Lazaro-Quintela M, Domine M, Vazquez Estevez S, Lopez-Vivanco G, Firvida Perez JL, Alonso Romero JL, Ferrera Delgado L, Garcia Giron C, Diz Tain P, Alvarez Alvarez R, Mut Sanchis P, Fernandez Canton I, Manrique Abos I, Martinez Aguillo M, Gomez-Aldaravi Gutierrez L, Ortega Granados AL, Alvarez Cabellos R, Garcia Sebastian A, Garcia Sifuentes LF, Reguart N. Identification of ALK-positive patients with advanced NSCLC and real-world clinical experience with crizotinib in Spain (IDEALK study). Lung Cancer. 2022 Nov;173:83-93. doi: 10.1016/j.lungcan.2022.09.010. Epub 2022 Sep 19. PMID 36162227
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081057

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with advanced/metastatic non-small cell lung cancer (NSCLC) were recruited in this multicentre, observational post-authorisation study. Participants were included in 3 sub-studies: ALK incidence, ALK treatment and ROS1 treatment sub-study. A total of 692 participants were enrolled in the study (ALK incidence sub-study= 572, ALK treatment sub-study=70 participants excluding 21 participants who were included from ALK incidence sub-study and ROS1 sub-study: 50).
Groups:
- ALK Incidence Sub-study: All participants with advanced/metastatic Non-Small Cell Lung Cancer (NSCLC) diagnosed at the hospital and who underwent Anaplastic Lymphoma Kinase (ALK) translocation molecular testing subsequently were included in the incidence sub-study.
- ALK Treatment Sub-study: Participants with advanced/metastatic NSCLC with confirmed ALK-positive translocation and who were treated with crizotinib in routine clinical practice retrospectively from January 2014 or prospectively during the study were included.
- ROS1 Treatment Sub-study: Participants with advanced/metastatic NSCLC with confirmed ROS1-positive translocation and who were treated with crizotinib in routine clinical practice on or after 08-Feb-2017 were included.
Period: ALK Incidence Sub-study
Arm/Group | ALK Incidence Sub-study | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Started | 572 | 0 | 0
Full Analysis Set | 559 | 0 | 0
Safety Analysis Set | 0 | 0 | 0
Completed | 572 | 0 | 0
Not Completed | 0 | 0 | 0
Period: ALK Treatment Sub-study
Arm/Group | ALK Incidence Sub-study | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Started | 0 | 91 (21 participants were included from ALK Incidence sub-study) | 0
Full Analysis Set | 0 | 91 | 0
Safety Analysis Set | 0 | 91 | 0
Completed | 0 | 91 | 0
Not Completed | 0 | 0 | 0
Period: ROS1 Treatment Sub-study
Arm/Group | ALK Incidence Sub-study | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Started | 0 | 0 | 50
Full Analysis Set | 0 | 0 | 50
Safety Analysis Set | 0 | 0 | 50
Completed | 0 | 0 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: ALK incidence sub-study- analysis population included all participants who presented an evaluable test for ALK translocation. ALK treatment sub-study- analysis population included only those participants exclusive to ALK treatment sub-study with confirmed ALK-positive translocation & who received treatment with crizotinib. ROS1 treatment sub-study- analysis population included all participants who had confirmed ROS1 translocation and had received atleast 1 dose of crizotinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALK Incidence Sub-study | ALK Treatment Sub-study | ROS1 Treatment Sub-study | Total
Number analyzed (Participants) | 559 | 70 | 50 | 679
Age, Customized [Count of Participants; unit: Participants]
  20 to 90 years | 559 | 70 | 50 | 679
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 45 | 28 | 268
  Male | 364 | 25 | 22 | 411
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and ethnicity were not collected. Population: Race and Ethnicity were not collected from any participant.
Number of Participants Classified According to Smoking Status [Count of Participants; unit: Participants] — Number for participants classified according to smoking status (non-smoker, former smoker, smoker) were reported in this baseline characteristic.
  Participants
    Non-smoker | 89 | 38 | 24 | 151
    Former-smoker | 256 | 17 | 17 | 290
    Smoker | 214 | 15 | 9 | 238
Previous Relevant Medical History: ALK Treatment Sub-study and ROS1 Sub-study [Count of Participants; unit: Participants] — Number of participants according to previous medical history were reported in this baseline characteristic. One participant may have more than one previous medical history. Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    Cardiovascular disease: number analyzed (Participants) | 0 | 70 | 50 | 120
    Cardiovascular disease | 0 | 18 | 35 | 53
    Neoplasm diseases: number analyzed (Participants) | 0 | 70 | 50 | 120
    Neoplasm diseases | 0 | 6 | 10 | 16
    Gastrointestinal disorders: number analyzed (Participants) | 0 | 70 | 50 | 120
    Gastrointestinal disorders | 0 | 6 | 6 | 12
    Pulmonary diseases: number analyzed (Participants) | 0 | 70 | 50 | 120
    Pulmonary diseases | 0 | 4 | 4 | 8
    Surgery: number analyzed (Participants) | 0 | 70 | 50 | 120
    Surgery | 0 | 23 | 22 | 45
    Other: number analyzed (Participants) | 0 | 70 | 50 | 120
    Other | 0 | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Eastern Cooperative Oncology Group (ECOG) Quality of Life Score: ALK Treatment and ROS1 Sub-study Only
Description: ECOG quality of life score is a rating of a participant's disease status, daily living activities and quality of life, where 0: fully active, 1: restricted in physically strenuous activity, 2: ambulatory and capable of self-care but unable to work, 3: capable only of limited self-care , 4: completely disabled; cannot carry on any self-care; totally confined to bed or chair, 5: dead. Higher scores indicated more severe disease, difficulty in performing daily activity and poor quality of life. Number of participants classified according to ECOG quality of life scores were reported in this outcome measure.
Time Frame: At baseline (for ALK treatment sub-study: at the beginning of diagnosis of ALK; for ROS1 treatment sub-study: at the beginning of diagnosis of ROS1 metastatic disease)
Population: ALK treatment sub-study: analysis population included all participants with confirmed ALK-positive translocation and who received treatment with crizotinib. ROS1 treatment sub-study: analysis population included all participants who had confirmed ROS1 translocation and had received at least 1 dose of crizotinib. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 81 | 42
Participants
  0 | 35 | 11
  1 | 43 | 29
  2 | 2 | 2
  3 | 1 | 0
  4 | 0 | 0
  5 | 0 | 0

2. Primary Outcome: Number of Participants Classified According to the Origin of Tumor Sample
Description: Number of participants classified according to the origin of tumor sample (primary tumor or metastasis) were reported in this outcome measure.
Time Frame: At baseline (for ALK incidence sub-study: at the beginning of initial diagnosis of lung cancer; for ROS1 and ALK treatment sub-study: at the beginning of ALK and ROS1 initial diagnosis)
Population: For ALK incidence sub-study, analysis population included all participants who presented an evaluable test for ALK translocation. For ALK treatment sub-study, analysis population included all participants with confirmed ALK-positive translocation and who received treatment with crizotinib. For ROS1 treatment sub-study, analysis population included all participants who had confirmed ROS1 translocation and had received at least 1 dose of crizotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Incidence Sub-study | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 559 | 91 | 50
Participants
  Primary tumor | 409 | 63 | 28
  Metastases | 150 | 28 | 22

3. Primary Outcome: Number of Participants Classified According to Type of Sample Collected for Tumor Analysis
Description: Number of participants classified according to the type of sample collected (biopsy, cell block or cytology) were reported in this outcome measure.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Incidence Sub-study | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 559 | 91 | 50
Participants
  Biopsy | 466 | 75 | 40
  Cell Block | 27 | 1 | 5
  Cytology | 66 | 15 | 5

4. Primary Outcome: Number of Participants Classified According to Histological Subtype of Tumor
Description: Number of participants classified according to the histological subtype (adenocarcinoma, squamous, large cell, not otherwise specified [NOS], other) were reported in this outcome measure.
Time Frame: At baseline (for ALK incidence sub-study: at the beginning of initial diagnosis of lung cancer; for ROS1 and ALK treatment sub-study: at the beginning of diagnosis of ALK and ROS1 metastatic disease)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Incidence Sub-study | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 559 | 91 | 50
Participants
  Adenocarcinoma | 453 | 84 | 44
  Squamous | 71 | 1 | 2
  Large Cell | 19 | 3 | 1
  NOS | 16 | 2 | 3
  Other | 0 | 1 | 0

5. Primary Outcome: Number of Participants Classified According to Stage of Tumor: ALK Treatment Sub-study and ROS1 Treatment Sub-study
Description: Tumor Node Metastasis (TNM): based on tumor size, metastasis to nearby lymph nodes (LN), or distant metastasis. Stages were: stage IIIA (T0N2M0, T1N2M0,T2N3M0, T3N1 or N2M0), stage IIIB (T4 any NM0, any TN3M0), stage IV (any T any NM1), where T0 = early form of tumor, T1 = less than (<) 2 centimeter (cm), T2 = 2-5 cm, T3 = greater than (>) 5 cm, T4 = large sized, N0 = not spread to lymph nodes (LN), N1 = spread to 1 to 3 LN, N2 = spread to 4 to 9 LN, N3 = spread >10 axillary LN, M0 = no metastasis, M1 = metastasis. The number of participants classified according to stages of tumor (Stage IIIA, IIIB and IV) were reported in this outcome measure.
Time Frame: At baseline (for ALK incidence sub-study: at the beginning of initial diagnosis of lung cancer; for ROS1 and ALK treatment sub-study: at the beginning of ALK and ROS1 initial diagnosis of metastatic disease)
Population: ALK treatment sub-study: analysis population included all participants with confirmed ALK-positive translocation and who received treatment with crizotinib. ROS1 treatment sub-study: analysis population included all participants who had confirmed ROS1 translocation and had received at least 1 dose of crizotinib. This outcome measure was planned to be analyzed for ALK treatment sub-study and ROS1 treatment sub-study only.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 91 | 50
Participants
  Stage IIIA | 5 | 1
  Stage IIIB | 8 | 7
  Stage IV | 78 | 42

6. Primary Outcome: Number of Participants Classified According to Molecular Alterations in Tumor: ALK Treatment Sub-Study and ROS1 Treatment Sub-Study
Description: Number of participants classified according to molecular alterations (PD-L1+: programmed death-ligand 1 positive, MET+: mesenchymal epithelial transition factor receptor positive, TP53+: tumor protein 53 positive, AKT: serine/threonine-protein kinase) in tumors were reported in this outcome measure.
Time Frame: as for outcome 1
Population: ALK treatment sub-study: all participants with confirmed ALK-positive translocation and who received treatment with crizotinib.ROS1 treatment sub-study: all participants who had confirmed ROS1 translocation and had received at least 1 dose of crizotinib.Here,'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.This outcome measure was planned to be analyzed for ALK treatment sub-study and ROS1 treatment sub-study only.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 5 | 16
Participants
  PD-L1+ | 4 | 14
  TP53+ | 1 | 0
  AKT | 0 | 1
  MET | 0 | 1

7. Primary Outcome: Number of Participants Classified According to Location of Metastases: ALK Treatment Sub-Study and ROS1 Treatment Sub-Study
Description: Number of participants classified according to the location of metastases were reported in this outcome measure. One participant may have more than one site of metastases.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 91 | 50
Participants
  Lymph nodes | 30 | 16
  Lung/Pleura | 42 | 18
  Bone | 34 | 14
  Brain | 11 | 4
  Liver | 12 | 7
  Other | 14 | 22

8. Primary Outcome: Number of Participants Categorized According to Number of Treatments Prior to Crizotinib: ALK Treatment Sub-Study and ROS1 Treatment Sub-Study
Description: Number of participants classified according to number of treatments (1 or 2) prior to crizotinib were reported in this outcome measure.
Time Frame: At baseline (for ALK treatment sub-study: after initial diagnosis of ALK metastatic disease; for ROS1 treatment sub-study: after initial diagnosis of ROS1 metastatic disease)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 51 | 19
Participants
  1 prior treatment | 35 | 14
  2 prior treatments | 16 | 5

9. Primary Outcome: Number of Participants According to Treatment Response: ALK Treatment Sub-Study and ROS1 Treatment Sub-Study
Description: Number of participants with treatment response as complete response (CR): disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 millimeter [mm] short axis), partial response (PR): at least 30 percent (%) decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), progressive disease (PD): at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions were reported in this outcome measure.
Time Frame: From date of inclusion until last date of follow-up (ALK treatment sub-study: maximum of 96.5 months and ROS1 treatment sub-study: maximum of 46.6 months)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 91 | 50
Participants
  CR | 8 | 2
  PR | 40 | 20
  SD | 22 | 12
  PD | 11 | 11
  Not specified/ Not evaluable | 9 | 2
  Unknown | 1 | 3

10. Primary Outcome: Number of Participants Classified According to Survival Data: ALK Treatment Sub-Study and ROS1 Treatment Sub-Study
Description: The number of participants classified as dead or alive were reported in this outcome measure.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 91 | 50
Participants
  Dead | 38 | 25
  Alive | 53 | 25

11. Primary Outcome: Percentage of Participants With European Organization For Research And Treatment Of Cancer Quality Of Life Questionnaire (EORTC QLQ-C30) Scores: ALK Treatment Sub-study
Description: QLQ-C30: 30 item questionnaire consisted of a global health (GH) score, 5 functional domains, 8 symptom scales and single item about financial difficulties. All items were graded by severity experienced during previous week and used a 4-point-scale (1: not at all, 2: a little, 3: quite a bit, 4: very much). The scores were converted to health-related quality of life (HRQoL) scale ranging from 0 - 100. Higher GH and functional domain scores indicated better function and lower scores in symptom scales and single item indicated more severity. Positive changes from baseline indicated improvement and negative changes from baseline indicated worsening for GH and functional domains. Negative changes from baseline indicated improvement and higher levels of functioning and positive changes from baseline indicated worsening for symptom scale and single item. Stable indicated that the symptoms were neither improving nor worsening.
Time Frame: Baseline, End (day 28) of Cycles 1 and 3, and end of treatment (up to approximately 15.2 months)
Population: Analysis population included all participants with confirmed ALK-positive translocation and who received treatment with crizotinib. This outcome measure was planned to be analyzed in ALK treatment sub-study only. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' indicates number of participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study
Number analyzed (Participants) | 42
Participants
  Baseline-End cycle 1, Global QoL: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Global QoL: Improvement | 8
  Baseline-End cycle 1, Global QoL: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Global QoL: Stable | 9
  Baseline-End cycle 1, Global QoL: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Global QoL: Worsening | 4
  Baseline-End cycle 1, Physical functioning: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Physical functioning: Improvement | 3
  Baseline-End cycle 1, Physical functioning: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Physical functioning: Stable | 10
  Baseline-End cycle 1, Physical functioning: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Physical functioning: Worsening | 10
  Baseline-End cycle 1, Role functioning: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Role functioning: Improvement | 7
  Baseline-End cycle 1, Role functioning: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Role functioning: Stable | 8
  Baseline-End cycle 1, Role functioning: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Role functioning: Worsening | 8
  Baseline-End cycle 1, Emotional functioning: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Emotional functioning: Improvement | 4
  Baseline-End cycle 1, Emotional functioning: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Emotional functioning: Stable | 13
  Baseline-End cycle 1, Emotional functioning: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Emotional functioning: Worsening | 4
  Baseline-End cycle 1, Cognitive functioning: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Cognitive functioning: Improvement | 1
  Baseline-End cycle 1, Cognitive functioning: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Cognitive functioning: Stable | 13
  Baseline-End cycle 1, Cognitive functioning: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Cognitive functioning: Worsening | 7
  Baseline-End cycle 1, Social functioning: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Social functioning: Improvement | 4
  Baseline-End cycle 1, Social functioning: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Social functioning: Stable | 9
  Baseline-End cycle 1, Social functioning: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Social functioning: Worsening | 8
  Baseline-End cycle 1, Fatigue: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Fatigue: Improvement | 9
  Baseline-End cycle 1, Fatigue: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Fatigue: Stable | 6
  Baseline-End cycle 1, Fatigue: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Fatigue: Worsening | 8
  Baseline-End cycle 1, Nausea and vomiting: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Nausea and vomiting: Improvement | 8
  Baseline-End cycle 1, Nausea and vomiting: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Nausea and vomiting: Stable | 9
  Baseline-End cycle 1, Nausea and vomiting: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Nausea and vomiting: Worsening | 6
  Baseline-End cycle 1, Pain: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Pain: Improvement | 6
  Baseline-End cycle 1, Pain: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Pain: Stable | 10
  Baseline-End cycle 1, Pain: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Pain: Worsening | 7
  Baseline-End cycle 1, Dyspnoea: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dyspnoea: Improvement | 3
  Baseline-End cycle 1, Dyspnoea: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dyspnoea: Stable | 13
  Baseline-End cycle 1, Dyspnoea: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dyspnoea: Worsening | 7
  Baseline-End cycle 1, Insomnia: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Insomnia: Improvement | 5
  Baseline-End cycle 1, Insomnia: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Insomnia: Stable | 12
  Baseline-End cycle 1, Insomnia: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Insomnia: Worsening | 6
  Baseline-End cycle 1, Loss of appetite: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Loss of appetite: Improvement | 5
  Baseline-End cycle 1, Loss of appetite: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Loss of appetite: Stable | 14
  Baseline-End cycle 1, Loss of appetite: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Loss of appetite: Worsening | 4
  Baseline-End cycle 1, Constipation: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Constipation: Improvement | 6
  Baseline-End cycle 1, Constipation: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Constipation: Stable | 10
  Baseline-End cycle 1, Constipation: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Constipation: Worsening | 7
  Baseline-End cycle 1, Diarrhea: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Diarrhea: Improvement | 0
  Baseline-End cycle 1, Diarrhea: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Diarrhea: Stable | 14
  Baseline-End cycle 1, Diarrhea: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Diarrhea: Worsening | 7
  Baseline-End cycle 1, Economic difficulties: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Economic difficulties: Improvement | 3
  Baseline-End cycle 1, Economic difficulties: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Economic difficulties: Stable | 12
  Baseline-End cycle 1, Economic difficulties: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Economic difficulties: Worsening | 6
  Baseline-End cycle 3, Global QoL: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Global QoL: Improvement | 6
  Baseline-End cycle 3, Global QoL: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Global QoL: Stable | 7
  Baseline-End cycle 3, Global QoL: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Global QoL: Worsening | 4
  Baseline-End cycle 3, Physical functioning: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Physical functioning: Improvement | 1
  Baseline-End cycle 3, Physical functioning: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Physical functioning: Stable | 10
  Baseline-End cycle 3, Physical functioning: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Physical functioning: Worsening | 6
  Baseline-End cycle 3, Role functioning: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Role functioning: Improvement | 5
  Baseline-End cycle 3, Role functioning: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Role functioning: Stable | 7
  Baseline-End cycle 3, Role functioning: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Role functioning: Worsening | 4
  Baseline-End cycle 3, Emotional functioning: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Emotional functioning: Improvement | 5
  Baseline-End cycle 3, Emotional functioning: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Emotional functioning: Stable | 7
  Baseline-End cycle 3, Emotional functioning: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Emotional functioning: Worsening | 5
  Baseline-End cycle 3, Cognitive functioning: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Cognitive functioning: Improvement | 2
  Baseline-End cycle 3, Cognitive functioning: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Cognitive functioning: Stable | 8
  Baseline-End cycle 3, Cognitive functioning: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Cognitive functioning: Worsening | 7
  Baseline-End cycle 3, Social functioning: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Social functioning: Improvement | 3
  Baseline-End cycle 3, Social functioning: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Social functioning: Stable | 9
  Baseline-End cycle 3, Social functioning: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Social functioning: Worsening | 5
  Baseline-End cycle 3, Fatigue: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Fatigue: Improvement | 6
  Baseline-End cycle 3, Fatigue: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Fatigue: Stable | 6
  Baseline-End cycle 3, Fatigue: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Fatigue: Worsening | 5
  Baseline-End cycle 3, Nausea and vomiting: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Nausea and vomiting: Improvement | 4
  Baseline-End cycle 3, Nausea and vomiting: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Nausea and vomiting: Stable | 10
  Baseline-End cycle 3, Nausea and vomiting: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Nausea and vomiting: Worsening | 3
  Baseline-End cycle 3, Pain: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Pain: Improvement | 4
  Baseline-End cycle 3, Pain: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Pain: Stable | 7
  Baseline-End cycle 3, Pain: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Pain: Worsening | 6
  Baseline-End cycle 3, Dyspnoea: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Dyspnoea: Improvement | 3
  Baseline-End cycle 3, Dyspnoea: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Dyspnoea: Stable | 7
  Baseline-End cycle 3, Dyspnoea: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Dyspnoea: Worsening | 7
  Baseline-End cycle 3, Insomnia: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Insomnia: Improvement | 6
  Baseline-End cycle 3, Insomnia: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Insomnia: Stable | 7
  Baseline-End cycle 3, Insomnia: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Insomnia: Worsening | 4
  Baseline-End cycle 3, Loss of appetite: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Loss of appetite: Improvement | 5
  Baseline-End cycle 3, Loss of appetite: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Loss of appetite: Stable | 9
  Baseline-End cycle 3, Loss of appetite: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Loss of appetite: Worsening | 3
  Baseline-End cycle 3, Constipation: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Constipation: Improvement | 3
  Baseline-End cycle 3, Constipation: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Constipation: Stable | 9
  Baseline-End cycle 3, Constipation: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Constipation: Worsening | 5
  Baseline-End cycle 3, Diarrhea: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Diarrhea: Improvement | 0
  Baseline-End cycle 3, Diarrhea: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Diarrhea: Stable | 14
  Baseline-End cycle 3, Diarrhea: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Diarrhea: Worsening | 3
  Baseline-End cycle 3, Economic difficulties: Improvement: number analyzed (Participants) | 17
  Baseline-End cycle 3, Economic difficulties: Improvement | 3
  Baseline-End cycle 3, Economic difficulties: Stable: number analyzed (Participants) | 17
  Baseline-End cycle 3, Economic difficulties: Stable | 12
  Baseline-End cycle 3, Economic difficulties: Worsening: number analyzed (Participants) | 17
  Baseline-End cycle 3, Economic difficulties: Worsening | 2
  Baseline-End of treatment, Global QoL: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Global QoL: Improvement | 1
  Baseline-End of treatment, Global QoL: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Global QoL: Stable | 1
  Baseline-End of treatment, Global QoL: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Global QoL: Worsening | 2
  Baseline-End of treatment, Physical functioning: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Physical functioning: Improvement | 0
  Baseline-End of treatment, Physical functioning: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Physical functioning: Stable | 3
  Baseline-End of treatment, Physical functioning: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Physical functioning: Worsening | 2
  Baseline-End of treatment, Role functioning: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Role functioning: Improvement | 1
  Baseline-End of treatment, Role functioning: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Role functioning: Stable | 1
  Baseline-End of treatment, Role functioning: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Role functioning: Worsening | 3
  Baseline-End of treatment, Emotional functioning: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Emotional functioning: Improvement | 0
  Baseline-End of treatment, Emotional functioning: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Emotional functioning: Stable | 2
  Baseline-End of treatment, Emotional functioning: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Emotional functioning: Worsening | 2
  Baseline-End of treatment, Cognitive functioning: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Cognitive functioning: Improvement | 1
  Baseline-End of treatment, Cognitive functioning: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Cognitive functioning: Stable | 3
  Baseline-End of treatment, Cognitive functioning: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Cognitive functioning: Worsening | 0
  Baseline-End of treatment, Social functioning: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Social functioning: Improvement | 0
  Baseline-End of treatment, Social functioning: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Social functioning: Stable | 3
  Baseline-End of treatment, Social functioning: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Social functioning: Worsening | 1
  Baseline-End of treatment, Fatigue: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Fatigue: Improvement | 2
  Baseline-End of treatment, Fatigue: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Fatigue: Stable | 0
  Baseline-End of treatment, Fatigue: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Fatigue: Worsening | 3
  Baseline-End of treatment, Nausea and vomiting: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Nausea and vomiting: Improvement | 1
  Baseline-End of treatment, Nausea and vomiting: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Nausea and vomiting: Stable | 3
  Baseline-End of treatment, Nausea and vomiting: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Nausea and vomiting: Worsening | 1
  Baseline-End of treatment, Pain: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Pain: Improvement | 2
  Baseline-End of treatment, Pain: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Pain: Stable | 0
  Baseline-End of treatment, Pain: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Pain: Worsening | 3
  Baseline-End of treatment, Dyspnoea: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Dyspnoea: Improvement | 0
  Baseline-End of treatment, Dyspnoea: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Dyspnoea: Stable | 3
  Baseline-End of treatment, Dyspnoea: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Dyspnoea: Worsening | 2
  Baseline-End of treatment, Insomnia: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Insomnia: Improvement | 2
  Baseline-End of treatment, Insomnia: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Insomnia: Stable | 1
  Baseline-End of treatment, Insomnia: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Insomnia: Worsening | 2
  Baseline-End of treatment, Loss of appetite: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Loss of appetite: Improvement | 1
  Baseline-End of treatment, Loss of appetite: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Loss of appetite: Stable | 2
  Baseline-End of treatment, Loss of appetite: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Loss of appetite: Worsening | 2
  Baseline-End of treatment, Constipation: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Constipation: Improvement | 1
  Baseline-End of treatment, Constipation: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Constipation: Stable | 3
  Baseline-End of treatment, Constipation: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Constipation: Worsening | 1
  Baseline-End of treatment, Diarrhea: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Diarrhea: Improvement | 0
  Baseline-End of treatment, Diarrhea: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Diarrhea: Stable | 3
  Baseline-End of treatment, Diarrhea: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Diarrhea: Worsening | 1
  Baseline-End of treatment, Economic difficulties: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Economic difficulties: Improvement | 0
  Baseline-End of treatment, Economic difficulties: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Economic difficulties: Stable | 2
  Baseline-End of treatment, Economic difficulties: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Economic difficulties: Worsening | 2

12. Primary Outcome: Percentage of Participants With European Organization For Research And Treatment Of Cancer Quality Of Life Questionnaire-Lung Cancer 13 (EORTC QLQ-LC13) Scores: ALK Treatment Sub-study
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer & treatment side effects typical of treatment with chemotherapy and radiotherapy. It comprised of multi-item scale and single-item scale for symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, & medicine for pain). Response range - 1: Not at all to 4: Very much. The scores were converted to a HRQoL scale ranging from 0 - 100 where, higher scores = greater level of symptoms. Negative changes from baseline indicated improvement and positive changes from baseline indicated worsening. Stable indicated that the symptoms were neither improving nor deteriorating.
Time Frame: Baseline, End (day 28) of Cycles 1 and 3, and end of treatment (up to approximately 15.2 months)
Population: Analysis population included all participants with confirmed ALK-positive translocation and who received treatment with crizotinib. This outcome measure was planned to be analyzed for ALK treatment sub-study only. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' indicates number of participants evaluable at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study
Number analyzed (Participants) | 42
Participants
  Baseline-End cycle 1, Dyspnoea: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dyspnoea: Improvement | 5
  Baseline-End cycle 1, Dyspnoea: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dyspnoea: Stable | 9
  Baseline-End cycle 1, Dyspnoea: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dyspnoea: Worsening | 9
  Baseline-End cycle 1, Cough: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Cough: Improvement | 8
  Baseline-End cycle 1, Cough: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Cough: Stable | 11
  Baseline-End cycle 1, Cough: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Cough: Worsening | 5
  Baseline-End cycle 1, Hemoptysis: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Hemoptysis: Improvement | 1
  Baseline-End cycle 1, Hemoptysis: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Hemoptysis: Stable | 22
  Baseline-End cycle 1, Hemoptysis: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Hemoptysis: Worsening | 0
  Baseline-End cycle 1, Sore mouth: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Sore mouth: Improvement | 1
  Baseline-End cycle 1, Sore mouth: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Sore mouth: Stable | 21
  Baseline-End cycle 1, Sore mouth: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Sore mouth: Worsening | 0
  Baseline-End cycle 1, Dysphagia: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dysphagia: Improvement | 3
  Baseline-End cycle 1, Dysphagia: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dysphagia: Stable | 18
  Baseline-End cycle 1, Dysphagia: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Dysphagia: Worsening | 2
  Baseline-End cycle 1, Peripheral neuropathy: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Peripheral neuropathy: Improvement | 4
  Baseline-End cycle 1, Peripheral neuropathy: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Peripheral neuropathy: Stable | 14
  Baseline-End cycle 1, Peripheral neuropathy: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Peripheral neuropathy: Worsening | 5
  Baseline-End cycle 1, Alopecia: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Alopecia: Improvement | 2
  Baseline-End cycle 1, Alopecia: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Alopecia: Stable | 18
  Baseline-End cycle 1, Alopecia: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Alopecia: Worsening | 2
  Baseline-End cycle 1, Chest pain: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Chest pain: Improvement | 7
  Baseline-End cycle 1, Chest pain: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Chest pain: Stable | 13
  Baseline-End cycle 1, Chest pain: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Chest pain: Worsening | 3
  Baseline-End cycle 1, Arm/shoulder pain: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Arm/shoulder pain: Improvement | 9
  Baseline-End cycle 1, Arm/shoulder pain: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Arm/shoulder pain: Stable | 13
  Baseline-End cycle 1, Arm/shoulder pain: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Arm/shoulder pain: Worsening | 1
  Baseline-End cycle 1, Pain elsewhere: Improvement: number analyzed (Participants) | 23
  Baseline-End cycle 1, Pain elsewhere: Improvement | 7
  Baseline-End cycle 1, Pain elsewhere: Stable: number analyzed (Participants) | 23
  Baseline-End cycle 1, Pain elsewhere: Stable | 8
  Baseline-End cycle 1, Pain elsewhere: Worsening: number analyzed (Participants) | 23
  Baseline-End cycle 1, Pain elsewhere: Worsening | 6
  Baseline-End cycle 3, Dyspnoea: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Dyspnoea: Improvement | 3
  Baseline-End cycle 3, Dyspnoea: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Dyspnoea: Stable | 6
  Baseline-End cycle 3, Dyspnoea: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Dyspnoea: Worsening | 7
  Baseline-End cycle 3, Cough: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Cough: Improvement | 7
  Baseline-End cycle 3, Cough: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Cough: Stable | 6
  Baseline-End cycle 3, Cough: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Cough: Worsening | 3
  Baseline-End cycle 3, Hemoptysis: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Hemoptysis: Improvement | 0
  Baseline-End cycle 3, Hemoptysis: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Hemoptysis: Stable | 16
  Baseline-End cycle 3, Hemoptysis: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Hemoptysis: Worsening | 0
  Baseline-End cycle 3, Sore mouth: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Sore mouth: Improvement | 1
  Baseline-End cycle 3, Sore mouth: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Sore mouth: Stable | 14
  Baseline-End cycle 3, Sore mouth: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Sore mouth: Worsening | 1
  Baseline-End cycle 3, Dysphagia: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Dysphagia: Improvement | 4
  Baseline-End cycle 3, Dysphagia: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Dysphagia: Stable | 10
  Baseline-End cycle 3, Dysphagia: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Dysphagia: Worsening | 1
  Baseline-End cycle 3, Peripheral neuropathy: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Peripheral neuropathy: Improvement | 2
  Baseline-End cycle 3, Peripheral neuropathy: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Peripheral neuropathy: Stable | 8
  Baseline-End cycle 3, Peripheral neuropathy: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Peripheral neuropathy: Worsening | 6
  Baseline-End cycle 3, Alopecia: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Alopecia: Improvement | 4
  Baseline-End cycle 3, Alopecia: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Alopecia: Stable | 11
  Baseline-End cycle 3, Alopecia: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Alopecia: Worsening | 0
  Baseline-End cycle 3, Chest pain: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Chest pain: Improvement | 2
  Baseline-End cycle 3, Chest pain: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Chest pain: Stable | 10
  Baseline-End cycle 3, Chest pain: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Chest pain: Worsening | 4
  Baseline-End cycle 3, Arm/shoulder pain: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Arm/shoulder pain: Improvement | 5
  Baseline-End cycle 3, Arm/shoulder pain: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Arm/shoulder pain: Stable | 10
  Baseline-End cycle 3, Arm/shoulder pain: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Arm/shoulder pain: Worsening | 0
  Baseline-End cycle 3, Pain elsewhere: Improvement: number analyzed (Participants) | 16
  Baseline-End cycle 3, Pain elsewhere: Improvement | 3
  Baseline-End cycle 3, Pain elsewhere: Stable: number analyzed (Participants) | 16
  Baseline-End cycle 3, Pain elsewhere: Stable | 8
  Baseline-End cycle 3, Pain elsewhere: Worsening: number analyzed (Participants) | 16
  Baseline-End cycle 3, Pain elsewhere: Worsening | 3
  Baseline-End of treatment, Dyspnoea: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Dyspnoea: Improvement | 1
  Baseline-End of treatment, Dyspnoea: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Dyspnoea: Stable | 0
  Baseline-End of treatment, Dyspnoea: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Dyspnoea: Worsening | 4
  Baseline-End of treatment, Cough: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Cough: Improvement | 4
  Baseline-End of treatment, Cough: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Cough: Stable | 1
  Baseline-End of treatment, Cough: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Cough: Worsening | 0
  Baseline-End of treatment, Hemoptysis: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Hemoptysis: Improvement | 0
  Baseline-End of treatment, Hemoptysis: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Hemoptysis: Stable | 5
  Baseline-End of treatment, Hemoptysis: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Hemoptysis: Worsening | 0
  Baseline-End of treatment, Sore mouth: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Sore mouth: Improvement | 0
  Baseline-End of treatment, Sore mouth: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Sore mouth: Stable | 5
  Baseline-End of treatment, Sore mouth: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Sore mouth: Worsening | 0
  Baseline-End of treatment, Dysphagia: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Dysphagia: Improvement | 1
  Baseline-End of treatment, Dysphagia: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Dysphagia: Stable | 4
  Baseline-End of treatment, Dysphagia: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Dysphagia: Worsening | 0
  Baseline-End of treatment, Peripheral neuropathy: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Peripheral neuropathy: Improvement | 0
  Baseline-End of treatment, Peripheral neuropathy: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Peripheral neuropathy: Stable | 3
  Baseline-End of treatment, Peripheral neuropathy: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Peripheral neuropathy: Worsening | 2
  Baseline-End of treatment, Alopecia: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Alopecia: Improvement | 0
  Baseline-End of treatment, Alopecia: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Alopecia: Stable | 5
  Baseline-End of treatment, Alopecia: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Alopecia: Worsening | 0
  Baseline-End of treatment, Chest pain: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Chest pain: Improvement | 1
  Baseline-End of treatment, Chest pain: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Chest pain: Stable | 4
  Baseline-End of treatment, Chest pain: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Chest pain: Worsening | 0
  Baseline-End of treatment, Arm/shoulder pain: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Arm/shoulder pain: Improvement | 2
  Baseline-End of treatment, Arm/shoulder pain: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Arm/shoulder pain: Stable | 3
  Baseline-End of treatment, Arm/shoulder pain: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Arm/shoulder pain: Worsening | 0
  Baseline-End of treatment, Pain elsewhere: Improvement: number analyzed (Participants) | 5
  Baseline-End of treatment, Pain elsewhere: Improvement | 1
  Baseline-End of treatment, Pain elsewhere: Stable: number analyzed (Participants) | 5
  Baseline-End of treatment, Pain elsewhere: Stable | 2
  Baseline-End of treatment, Pain elsewhere: Worsening: number analyzed (Participants) | 5
  Baseline-End of treatment, Pain elsewhere: Worsening | 2

13. Primary Outcome: Percentage of Participants With Anaplastic Lymphoma Kinase Positive Translocations: ALK Incidence Sub-Study
Description: The percentage of participants with ALK positive translocations were reported in this outcome measure.
Time Frame: At baseline (after initial diagnosis of lung cancer and until end of recruitment of ALK incidence sub study)
Population: Analysis population included all participants presented an evaluable test for ALK translocation. This outcome measure was planned to be analyzed for ALK incidence sub-study only.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Incidence Sub-study
Number analyzed (Participants) | 559
Participants | 31

14. Primary Outcome: Progression-Free Survival (PFS): ALK Treatment Sub-study and ROS1 Treatment Sub-Study
Description: Progression-free survival (PFS) was defined as the period between the first day of treatment and the first day that progressive disease (PD) (at least a 20% increase [including an absolute increase of at least 5 mm] in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions) was observed according to response evaluation criteria in solid tumors (RECIST) criteria, or death. Participants who have not had an event at the time of the analysis of the study data were censored at the date of the last available follow-up.
Time Frame: From first day of treatment until date of progressive disease, death or censored, whichever was the earliest (ALK treatment sub-study: maximum of 96.5 months and ROS1 treatment sub-study: maximum of 46.6 months)
Population: For ALK treatment sub-study, analysis population included all participants with confirmed ALK-positive translocation and who received treatment with crizotinib. For ROS1 treatment sub-study, analysis population included all participants who had confirmed ROS1 translocation and had received at least 1 dose of crizotinib. This outcome measure was planned to be analyzed for ALK treatment sub-study and ROS1 treatment sub-study only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 91 | 50
Months | 15.8 [11.8 to 22.3] | 7.5 [4.0 to 10.1]

15. Primary Outcome: Objective Response Rate (ORR): ALK Treatment Sub-study and ROS1 Treatment Sub-Study
Description: ORR: percentage of participants who achieved CR : disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size(<10 mm short axis), or PR : at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Additionally, the participants with SD : neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, PD: at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions were evaluated. The participants were evaluated in accordance with RECIST criteria.
Time Frame: From first day of treatment until date of CR, PR or SD (ALK treatment sub-study: maximum of 96.5 months and ROS1 treatment sub-study: maximum of 46.6 months)
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 81 | 45
Percentage of participants | 59.3 | 48.9

16. Primary Outcome: Duration of Response (DOR): ALK Treatment Sub-study and ROS1 Sub-Study
Description: Duration of response (DOR) in participants with PR or CR was defined as the interval from the date the best response was documented to the first date that progressive disease (at least a 20% increase [including an absolute increase of at least 5 mm] in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions) was observed.
Time Frame: From the date the best response was documented until the date of progressive disease (ALK treatment sub-study: maximum of 96.5 months and ROS1 treatment sub-study: maximum of 46.6 months)
Population: as for outcome 6
Measure: Median (Full Range); unit: Months
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 32 | 16
Months | 13.5 [0.0 to 48.3] | 4.4 [0.0 to 25.2]

17. Primary Outcome: Overall Survival (OS): ALK Treatment Sub-study and ROS1 Treatment Sub-Study
Description: Overall survival (OS) was defined as the period from the first day of treatment until death or censored up to the last date on which it was known that the participant was alive.
Time Frame: From first day of treatment until date of death or censored, whichever was earliest (ALK treatment sub-study: maximum of 96.5 months and ROS1 treatment sub-study: maximum of 46.6 months)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 91 | 50
Months | 46.5 [34.6 to NA] — Upper limit of 95% CI could not be calculated due to a smaller number of participants with event. | 21.9 [9.8 to NA] — Upper limit of 95% CI could not be calculated due to a smaller number of participants with event.

18. Primary Outcome: Number of Participants With Adverse Events According to Seriousness: ALK Treatment Sub-study and ROS1 Treatment Sub-Study
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. SAE was defined as any untoward medical occurrence at any dose that: resulted in death, was life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was important medical event; required hospitalization or prolongation of existing hospitalization. The number of participants with non-SAEs and SAEs were reported in this outcome measure.
Time Frame: From start of study treatment until end of follow-up (ALK treatment sub-study: maximum of 96.5 months and ROS1 treatment sub-study: maximum of 46.6 months)
Population: Safety population included all participants with advanced/metastatic NSCLC with confirmed ALK/ROS1 positive translocation who met all the study screening criteria and had received at least one dose of treatment with crizotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
Number analyzed (Participants) | 91 | 50
Participants
  Non-SAEs | 54 | 33
  SAEs | 25 | 9

ADVERSE EVENTS:
Time Frame: From start of study treatment until end of follow-up (ALK treatment sub-study: maximum of 96.5 months and ROS1 treatment sub-study: maximum of 46.6 months)
Description: An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both serious and non-serious event. Safety population: analysis included participants with advanced/metastatic NSCLC with confirmed ALK/ROS1 positive translocation who met all study screening criteria and had at least 1 dose of crizotinib treatment. Data was not collected for ALK Incidence sub-study as the pre-defined criteria for safety collection did not meet.
Arm/Group | ALK Treatment Sub-study | ROS1 Treatment Sub-study
All-Cause Mortality (participants affected / at risk) | 38/91 | 25/50
Serious Adverse Events (participants affected / at risk) | 25/91 | 9/50
Other Adverse Events (participants affected / at risk) | 54/91 | 33/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALK Treatment Sub-study (N=91) | ROS1 Treatment Sub-study (N=50)
Transaminases increased (Investigations) | 6 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
General deterioration of physical condition (General disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post-intervention complication (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALK Treatment Sub-study (N=91) | ROS1 Treatment Sub-study (N=50)
Elevated alanine aminotransferase (Investigations) | 8 | 7
Elevated amylase (Investigations) | 1 | 0
Elevated aspartate aminotransferase (Investigations) | 6 | 7
Increased blood alkaline phosphatase (Investigations) | 1 | 0
Elevated Gamma glutamyl transferase (Investigations) | 1 | 0
Increased QT Interval electrocardiography (Investigations) | 1 | 0
Elevated Transaminases (Investigations) | 1 | 0
Decreased weight (Investigations) | 0 | 1
Oesophagic candidiasis (Infections and infestations) | 1 | 0
Candidiasis infection (Infections and infestations) | 1 | 0
Tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bradycardia (Cardiac disorders) | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 8 | 3
Amenorrhea (Reproductive system and breast disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Peripheric neurophathy (Nervous system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 13 | 7
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Upper abdominal pain (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 10 | 3
Gastritis (Gastrointestinal disorders) | 1 | 0
Nauseous (Gastrointestinal disorders) | 15 | 8
Odynophagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 13 | 10
Oedema (General disorders) | 15 | 14
Pyrexia (General disorders) | 1 | 1
Hot flushes (General disorders) | 0 | 1
Vision disorders (Eye disorders) | 10 | 6
Photopsia (Eye disorders) | 2 | 0
Blepharitis/Meibomytis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Kidney impairment (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Effort dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT02679170/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT02679170/SAP_001.pdf